CLINICAL TRIAL: NCT03936894
Title: A Single Escalating Dose Pilot Trial of Canakinumab (ILARIS®) Assessing Safety and Biomarker Changes in Boys With Duchenne Muscular Dystrophy
Brief Title: Single Escalating Dose Pilot Trial of Canakinumab (ILARIS®) in Duchenne Muscular Dystrophy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's National Research Institute (Other)
Collaborators: Foundation to Eradicate Duchenne (Unknown)
Responsible Party: Principal Investigator, Christopher Spurney, Professor, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10234
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Canakinumab; Biomarker
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — canakinumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, single ascending dose pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Canakinumab treatment
  Interventions: Drug: Canakinumab Injection [Ilaris]

INTERVENTIONS:
Drug: Canakinumab Injection [Ilaris] — Subject receives subcutaneous injection of canakinumab 2 mg/ kg or 4 mg/kg

SUMMARY:
Canakinumab is an anti-interleukin 1 beta (IL1β) antibody approved for use in young children with familial Mediterranean fever, systemic onset juvenile idiopathic arthritis and TNF-receptor associated periodic fever syndrome. This study is a pilot trial to investigate the effects of canakinumab on clinical safety and potential clinical efficacy as demonstrated by short-term changes in select serum biomarkers in a sample of young boys with DMD who are most likely to have high levels of muscle inflammation. Steroid naive DMD subjects aged greater than or equal to 2 years old to less than 6 years old will receive a single subcutaneous dose of canakinumab and undergo safety and serum biomarker monitoring for 30 days. The first 3 subjects will receive 2 mg/kg and if well tolerated, the second 3 subjects will receive 4 mg/kg.

DETAILED DESCRIPTION:
The study is an open-label, single ascending dose study to assess safety and to evaluate short-term changes in biomarkers. The first 3 boys will receive canakinumab at a dose of 2 mg/kg, and the second 3 will receive a dose of 4 mg/kg. The study is comprised of four visits: a screening visit with baseline lab assessment, treatment day, a 10-14 day post-treatment evaluation with safety labs, and a 30 day post-treatment evaluation with safety labs. There will be a phone assessment on day 3-5 after treatment to screen for any side effects.

Clinical evaluation will screen for clinical AEs and SAEs. If dose escalation (4 mg/kg) must be terminated due to dose-limiting toxicities, the remaining subjects may be enrolled to evaluate the safety of canakinumab at the lower dose level (2 mg/kg).

One blood draw will occur after consent at least 48 hours prior to treatment day and on days 10-14 and 30 after the canakinumab injection to screen for laboratory abnormalities and collect serum for biomarker analysis. After obtaining consent, prior to treatment, 2 red top and 1 purple top 4 cc tubes will be obtained for screening labs and serum biomarker collection. Tuberculosis screening (Quantiferon-Gold) will use 4 blood tubes (grey, yellow, purple, green) with 1 cc of blood in each. At the following 2 visits with blood draws, two red top and one purple top collection tubes of 4 cc will be collected per subject. For red top blood collection tubes, one tube will be sent to the clinical lab for safety lab processing. The second tube will be processed in the research lab for serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent or legal guardian has provided written informed consent/HIPAA authorization prior to any study-related procedure
* Subject has a diagnosis of DMD
* Subject is ≥ 2 years of age at time of enrollment in the study
* Subject is naïve to treatment with glucocorticoids for DMD
* Subject is ambulatory
* Clinical laboratory test results are within the normal range at the Screening Visit, or if abnormal, are not clinically significant (includes less than 5x normal for AST and ALT), in the opinion of the Investigator. TB serology is negative.
* Subject and parent/guardian are willing and able to comply with, drug administration plan, and follow up visits.

Exclusion Criteria:

* Subject is <2 years of age
* Subject has current or history of major renal or hepatic impairment, diabetes mellitus or immunosuppression;
* Subject has current or history of chronic systemic fungal or viral infections;
* Subject has had an acute illness within 4 weeks prior to the first dose of study medication;
* Subject received live vaccination within the previous month
* Subject has evidence of symptomatic cardiomyopathy [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
* Subject is currently being treated or has received previous treatment with oral glucocorticoids or other immunosuppressive agents [Notes: Past transient use of oral glucocorticoids or other oral immunosuppressive agents for indication other than DMD for no longer than 3 months cumulative, with last use at least 3 months prior to first dose of study medication, will be considered for eligibility on a case-by-case basis. Inhaled and/or topical glucocorticoids prescribed for an indication other than DMD are permitted but must be administered at stable dose for at least 3 months prior to study drug administration];
* Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
* Subject is currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to the start of study treatment; Note: Any parameter/test may be repeated at the Investigator's discretion during Screening to determine reproducibility. In addition, subjects may be rescreened if ineligible due to a transient condition which would prevent the subject from participating, such as an upper respiratory tract infection or injury.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only males with genetically confirmed Duchenne muscular dystrophy are eligible
Enrollment: 3 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Clinical adverse events | 2 weeks
  Monitor for changes in health status related to medication use
Laboratory adverse events | 2 weeks
  Monitor for changes in laboratory results related to medication use
Clinical adverse events | 4 weeks
  Monitor for changes in health status related to medication use
Laboratory adverse events | 4 weeks
  Monitor for changes in laboratory results related to medication use

SECONDARY OUTCOMES:
Changes in serum biomarkers of inflammation after treatment | 2 weeks
  Monitor serum biomarker changes associated with anti-inflammatory properties including CD23, Protein C, CCL22, lymphotoxin a1/b1, CD49a, Ly9 and MMP-9, 12 and compare to baseline levels to demonstrate increase or decrease in biomarker levels
Changes in serum biomarkers of inflammation after treatment | 4 weeks
  Monitor serum biomarker changes associated with anti-inflammatory properties including CD23, Protein C, CCL22, lymphotoxin a1/b1, CD49a, Ly9 and MMP-9, 12 and compare to baseline levels to demonstrate increase or decrease in biomarker levels

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Spurney, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No